CLINICAL TRIAL: NCT05729438
Title: Nutritional Assesment in Patients With Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: SUUMC Central Military Hospital Dr Carol Davila (Other)
Responsible Party: Principal Investigator, Bucurica Sandica, Principal Investigator, Head of Functional Exploring Laboratory, SUUMC Central Military Hospital Dr Carol Davila
Other Study IDs: 559
Record Dates: First submitted 2023-01-31; First posted 2023-02-15 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Amino Acids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: BCAA — status of nutrition evaluation after 3 months of BCAA
  Other Names: branched chain amino acids

SUMMARY:
This study aims to evaluated nutritional status in patiets with cirrhosis

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age >18, <75 years old
* hepatic cirrhosis diagnosis

Exclusion Criteria:

* refuse to participate/to give consent
* presence of musculo-skeletal disease previous diagnosed, neuropathic diseases, malignancy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients males and females with hepatic cirrhosis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
muscle mass change | 3 months
  muscle mass changes in DEXA or body composition measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Suumc, Bucharest, București - Sector1, Romania

IPD SHARING:
Plan to Share IPD: Undecided